CLINICAL TRIAL: NCT07190261
Title: A Single-arm Phase 2 Prospective Clinical Study of Enatumab in the Treatment of Relapsed/Refractory Warm Antibody Autoimmune Hemolytic Anemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bing Han (Other)
Responsible Party: Sponsor-Investigator, Bing Han, Peking Union Medical College Hospital, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCMA/CD3+--R/R wAIHA
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Hemolytic Anemia
Keywords: Autoimmune Hemolytic Anemia; Enatumab; Single-arm phase 2 prospective
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Enatumab treat (Experimental): The recommended subcutaneous injection dose of this product is as follows: an incremental dose of 12mg on day 1, an incremental dose of 32mg on day 4, an initial treatment dose of 38mg on day 8, and subsequent treatment doses of 38mg in weeks 4 and 6.
  Interventions: Drug: enatumab

INTERVENTIONS:
Drug: enatumab — The recommended subcutaneous injection dose of this product is as follows: an incremental dose of 12mg on day 1, an incremental dose of 32mg on day 4, an initial treatment dose of 38mg on day 8, and subsequent treatment doses of 38mg in weeks 4 and 6.

SUMMARY:
Glucocorticoids are the first-line treatment for wAIHA, but patients are prone to recurrence after dose reduction or discontinuation of glucocorticoids. Birgens et al. 's study found that approximately 55% of patients treated with prednisolone monotherapy experienced recurrence at 36 months. The overall response rate of second-line treatment with rituximab is 70-80%, but the recurrence rate reaches 50%. The response rates of other immunosuppressants, such as cyclosporine, cyclophosphamide, and azathioprine, are relatively low, approximately 30-50%. Patients with chronic hemolysis have recurrent episodes, which affect their survival and quality of life. New treatment methods need to be explored.

DETAILED DESCRIPTION:
Enatumab (BCMA/CD3 bispecific antibody) is a bispecific T-cell articulation antibody targeting BCMA. Its Fab segment can bind to BCMA of plasma cells, plasma blasts and multiple myeloma cells as well as CD3 of T cells. It has shown good efficacy in the treatment of relapsed/refractory multiple myeloma (MM). Enatumab can specifically bind to BCMA on myeloma cells and CD3 on T cells. Through the production and release of cytokines, it activates T cells, promotes T cell proliferation, and releases cytotoxic molecules (including granzyme and perforin), thereby inducing apoptosis of myeloma cells. Plasma cells play a significant role in the pathogenesis of autoimmune diseases and are the main cells that produce autoantibodies. In AIHA, the production of autoantibodies is closely related to the abnormal activation and proliferation of plasma cells. These autoantibodies attack red blood cells, leading to hemolysis. Therefore, theoretically speaking, enatumab may improve the condition of patients with AIHA by inhibiting or eliminating abnormal plasma cells and reducing the production of autoantibodies. At present, there have been two reports internationally on the treatment of refractory AIHA with T-cell agonists targeting BCMA. In 2025, Shi Jun et al. reported two cases where BCAM-targeted T-cell agonists (CM336) successfully treated relapsed AIHA after chimeric antigen receptor T-cell (CAR-T) therapy targeting CD19. Patient 1 (a 10-year-old girl), with a 9-year history of Evans syndrome, still experienced recurrent hemolysis after multiple immunosuppressive treatments. Remission occurred within 14 days after the first CAR-T therapy, but recurred after 6.8 months. There was no response to the second CAR-T. Partial remission was achieved on the 13th day of CM336 treatment, and hemoglobin returned to normal on the 17th day. Case 2 (a 22-year-old female), with a 2-year history of AIHA, had no response to three immunosuppressants and splenectomy. She achieved remission within 10 days after CD19 CAR-T treatment and relapsed after 8.1 months. Partial remission was achieved on the 19th day of CM336 treatment, and hemoglobin returned to normal on the 21st day. The hemolytic indicators such as reticulocytes, LDH and indirect bilirubin in 2 patients decreased significantly and maintained remission for at least 6 months. The B cells and free light chains in the peripheral blood of the two patients decreased rapidly within 2 weeks after medication, and the B cells and plasma cells in the bone marrow were significantly cleared within 12 weeks. In terms of adverse reactions, Patient 1 developed grade 1 skin induration, and both patients presented with hypogammaglobulinemia. However, the overall safety was controllable. CM336 can effectively eliminate residual BCMA⁺ plasma cells, reverse the recurrence of multiple refractory AIHA after CAR-T, and provide a more targeted plasma cell-targeted immune strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender not limited.
2. Primary wAIHA with a clear diagnosis.
3. Patients who have relapsed or are refractory after at least second-line treatment (previous treatments include at least two types of glucocorticoids, CD20 monoclonal antibodies or other immunosuppressants). Refractory is defined as failure to achieve partial remission after 6 months of treatment with a stable dose of immunosuppressants.
4. The infusion of CD20 monoclonal antibody should be at least three months apart. If taking immunosuppressants such as cyclosporine and sirolimus, the medication should be discontinued for at least one month.
5. Hemoglobin (HGB) ≤100g/ and ≥ 60g/L.
6. Before treatment, the patient's alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were less than 3 times the upper limit of normal (ULN), and the serum creatinine was less than 1.5 times ULN.
7. Voluntarily join this study, sign the informed consent form with good compliance, and be willing to cooperate with regular follow-ups for efficacy evaluation and side effect monitoring.

Exclusion Criteria:

* (1) Those with impaired functions of organs such as the heart, liver and lungs; Patients with acute renal insufficiency.

  (2) Patients with connective tissue diseases and other secondary AIHA. (3) There is an active infection of hepatitis B virus (HBV), hepatitis C virus (HCV), severe acute respiratory syndrome coronavirus 2 (SARS-CoV2), human immunodeficiency virus (HIV), or any uncontrolled bacterial, fungal or viral infection.

  (4) Complicated with malignant tumors or a history of tumors. (5) When screening, the subjects had other types of uncorrected anemia, such as nutritional anemia, etc.

  (6) Had received other BCMA-targeted or CART treatments before screening. (7) Pregnant or lactating women. (8) Activity ≥ grade 2 peripheral sensory/motor neuropathy. (9) Had received treatment with other experimental drugs within 30 days (or as required by local regulations) or within 5 half-lives (whichever is longer) prior to the first use of the intervention drug in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2027-09-18 (Estimated); Study Completion 2027-09-18 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | 3 months
  The overall response rate (ORR) and complete response rate (CRR) at 3 months. The overall response rate (ORR) is defined as the ratio of patients achieving complete response (CR) plus partial response (PR)

SECONDARY OUTCOMES:
The incidence and severity of adverse events | 6-months
  Safety analyses include assessments of the incidence and severity of adverse events; all adverse events that occurred or worsened during the treatment period will be reported, as well as adverse events that occurred later but are considered by the investigator to be related to the trial drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Shuangfuyuan, NO I., China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data would be accepted upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10years
Access Criteria: email request